CLINICAL TRIAL: NCT06854874
Title: Validation Study of the Italian Version of the "Assessment of Life Habits 4.0" Scale (LIFE-H) for Measuring Participation in Children With Disabilities Aged 5 to 13 Years
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Silvia Paoli, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: LFH01
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Validation Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUNG In Italy there are still few translated and validated instruments to assess participation.

In the field of pediatric rehabilitation, among the tools available internationally, one of the most comprehensive and widely used is the Assessment of Life Habits, or LIFE-H, now in its 4.0 version. The LIFE-H scale was originally developed in French and implemented by the International Network on the Disability Creation Process - INDPC, also known as the Quebec Model or Handicap Creation Process.

Internationally, the "LIFE-H" scale has been translated and validated in several languages. The scale is among the most comprehensive and detailed instruments in the literature: it consists of 90 items (life habits), divided into 12 domains, 6 of which are for regular activities (e.g., communication and mobility), and 6 for social roles (responsibility and interpersonal relationships).

A study of Italian translation and cultural adaptation of the LIFE-H scale 4.0 for children aged 5 to 13 years, was carried out during 2020-2021.

The scale and its related user manual in Italian version have also been insert into the platform of the Canadian originator company "Réseau international sur le Processus de production du handicap" - RIPPH).

AIM The goal of the study is to assess the intra- and inter-rater reliability, internal consistency and construct validity of the scale in its Italian version.

METHOD Participants will be recruited from the pediatric rehabilitation centers of Toscana Centro , AOU Meyer IRCCS and AORN Santobono-Pausilipon Subjects interviewed will be caregivers of children with disabilities between the ages of 5 and 13 years. Care-givers of children with physical, sensory and cognitive disabilities, regardless of diagnosis, will be included in the study, as per the scale's user manual.

First Part Step 1: Presentation of the project through informational documentation to pediatric rehabilitation physical therapists of the territorial services of Toscana Centro and AOU Meyer IRCCS, who will identify candidate families for the study.

Step 2: Collection of informed consent by the investigating physical therapist in the referral area.

Step 3: TEST: Administration of the LIFE-H 4.0 / 5-13 years scale by an investigator (FT 1). As stipulated among the modes of administration, the questionnaire will be completed by the reference person or parent of the child with support from the experimenter. The administration will be done via video call on Google Meet platform, which platform is deemed most suitable in terms of use for families.

Step 4 : RETEST: After an interval of 15 days, second administration of the questionnaire will be carried out in the same manner and by the same experimenter.

Step 5 : Analysis and comparison of the collected data. Second part Step 6: Making contact with subjects who had adhered to both phases of the study (as indicated in the informed consent signed in step one) and re-enrollment through informational documentation to pediatric rehabilitation physical therapists from the territorial services of Toscana Centro, AOU Meyer IRCCS, and AORN Santobono-Pausilipon, who will identify candidate families for the study.

Step 7: Collection of informed consent from the investigating physical therapist in the target area.

Step 8: TEST: Administration of the LIFE-H 4.0 / 5-13 years scale by an investigator (FT 3). As stipulated among the modes of administration, the questionnaire will be completed by the reference person or parent of the child with support from the experimenter. The administration will be done via video call on Google Meet which platform is deemed most suitable in terms of family use.

Step 9: RETEST: Administration of the LIFE-H 4.0 / 5-13 years scale by an experimenter (FT 4) 15 days apart in the same manner.

Step 10: To complete the validation process (Construct Validity), the PEM-CY questionnaire will be provided to parents participating in the second phase of the study. The instrument was chosen, among the few available in the Italian language, because of features in common with the Life-H scale. The caregivers will be able to fill out the paper version of the questionnaire themselves. The latter will be kept within the child's medical record; the investigators will only be informed of the final score of the questionnaire.

step 11: analysis and comparison of collected data SAMPLE SIZING AND STATISTICAL METHODS OF DATA ANALYSIS With respect to the required sample size, contacts have been made with the Canadian authors of the LIFE-H scale (International Network on the Disability Creation Process - INDPC), who suggest a minimum minimum sample size of 30 subjects. Also taking into consideration other scale validation articles, we therefore plan to enroll 30 subjects for Phase 1 (intra-operator concordance and internal consistency) and 130 subjects for Phase 2 (inter-operator concordance and construct validity of construct). Analysis of the results of the LIFE-H questionnaire

ELIGIBILITY:
Inclusion Criteria:

* caregivers of children with physical, sensory, cognitive disabilities between the ages of 5 and 13 years.

Exclusion Criteria:

* Parents who do not master the Italian language
* Absence of signed informed consent from parents

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Caregivers of children with disabilities between the ages of 5 and 13 years. Care-givers of children with physical, sensory and cognitive disabilities, regardless of diagnosis, will be included in the study, as per the scale's user manual.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intra/inter-operator concordance (test-retest) will be estimated using the intraclass correlation coefficient (ICC) | Baseline and after 15 days
  Will consider poor scores between 0 and 0.20; fair between 0.21 and 0.40; moderate between 0, 41 and 0.60 ; good between 0.61 and 0.80; excellent between 0.81 and 1

SECONDARY OUTCOMES:
Internal consistency will be evaluated with Cronbach's Alph | Baseline and after 15 days
  A result ≥ of 0.7 will be considered relevant

OTHER OUTCOMES:
Construct validity will be assessed by r Rho | Baseline and after 15 days
  Will consider as strong correlation with r Rho ≥ 0.7

CONTACTS AND LOCATIONS:
Overall Officials: silvia paoli, pediatric Phisiotherapist MSc, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children Hospital IRCCS, Florence, Italy